CLINICAL TRIAL: NCT00210938
Title: A Multicenter, Double-Blind, Randomized, Phase 3 Study of Doripenem Versus Comparator Antibiotic in the Treatment of Complicated Intra-Abdominal Infections
Brief Title: Doripenem in the Treatment of Complicated Intra-Abdominal Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Peninsula Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005383
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Bacterial Infections and Mycoses; Appendicitis; Cholecystitis; Pancreatitis; Peritonitis
Keywords: Complicated Intra-Abdominal Infections; Appendicitis; Cholecystitis; Peritonitis
MeSH Terms: conditions — Bacterial Infections and Mycoses; Appendicitis; Cholecystitis; Pancreatitis; Peritonitis | interventions — Doripenem

INTERVENTIONS:
Drug: Doripenem

SUMMARY:
The purpose of this study is to compare the clinical response rates of doripenem versus a comparator antibiotic in treatment of hospitalized patients with complicated intra-abdominal infections.

DETAILED DESCRIPTION:
Doripenem is an antibiotic medication not yet approved by the US FDA. This is a phase 3, multicenter, prospective, randomized, double-blind study of intravenous doripenem versus a comparator antibiotic to assess the effectiveness and safety of doripenem in the treatment of complicated intra-abdominal infections in hospitalized adults. The primary endpoint is the clinical response rate measured at late follow-up visit. The patients will receive either doripenem or comparator; treatment duration is 5 to 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Has a requirement for surgical intervention within 24 hours of study entry
* Requirement of antibacterial therapy in addition to surgical intervention in certain intra-abdominal infections.

Exclusion Criteria:

* Female patients who are pregnant, nursing, or if of child bearing potential not using a medically accepted, effective method of birth control
* Any rapidly-progressing disease or immediately life-threatening illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2004-03; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Clinical response rate measured at late follow-up visit.

SECONDARY OUTCOMES:
Clinical response rate measured at early follow-up visit. Microbiological response rate at both early and late follow-up visits. Safety assessment (adverse events, changes in vital signs, laboratory tests results) conducted throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Kaniga K, Flamm R, Tong SY, Lee M, Friedland I, Redman R. Worldwide experience with the use of doripenem against extended-spectrum-beta-lactamase-producing and ciprofloxacin-resistant Enterobacteriaceae: analysis of six phase 3 clinical studies. Antimicrob Agents Chemother. 2010 May;54(5):2119-24. doi: 10.1128/AAC.01450-09. Epub 2010 Mar 8. PMID 20211892
- [Derived] Zhanel GG, Ketter N, Rubinstein E, Friedland I, Redman R. Overview of seizure-inducing potential of doripenem. Drug Saf. 2009;32(9):709-16. doi: 10.2165/00002018-200932090-00001. PMID 19670912
- See also: A Multicenter, Double-Blind, Randomized, Phase 3 Study to Compare the Safety and Efficacy of Intravenous Doripenem with that of Meropenem in Complicated Intra-abdominal Infections — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=637&filename=CR005383_CSR.pdf